CLINICAL TRIAL: NCT01431638
Title: A 36-week Open-label Extension Study of CACZ885H2361 on the Safety and Tolerability of Canakinumab 150 mg s.c. Pre-filled Syringe (PFS) in Treating Acute Gouty Arthritis Flares in Frequently Flaring Patients
Brief Title: Long-Term Safety and Tolerability of Canakinumab Prefilled Syringes in Frequently Flaring Acute Gouty Arthritis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885H2361E1; 2011-001342-15
Record Dates: First submitted 2011-08-30; First posted 2011-09-09 (Estimated); Results first posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-06

CONDITIONS: Acute Gouty Arthritis
Keywords: Gout; arthritis; gout flare; acute gout; gouty; rheumatic disease; uric acid; podagra
MeSH Terms: conditions — Gout; Arthritis; Rheumatic Diseases | interventions — canakinumab

STUDY DESIGN:
Intervention Model Description: Uncontrolled
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Canakinumab 150mg (Experimental): Canakinumab 150mg in prefilled syringe subcutaneously
  Interventions: Drug: Canakinumab 150mg in prefilled syringe

INTERVENTIONS:
Drug: Canakinumab 150mg in prefilled syringe — Canakinumab 150mg in prefilled syringe will be given in a single dose subcutaneously upon demand for gouty arthritis flares

SUMMARY:
This is a 36 week open-label extension of the canakinumab pre-filled syringe study for safety and tolerability in patients who have frequent flares of acute gouty arthritis.

ELIGIBILITY:
Inclusion criteria:

* Compliance and completion of the canakinumab PFS core study
* Unchanged significant clinical medical history from entry into core study

Exclusion criteria:

* Physician judgment of unsuitability for the study
* Pregnant or nursing women Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2011-08-25 (Actual); Primary Completion 2013-05-09 (Actual); Study Completion 2013-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (64):
- United States (53):
  - Novartis Investigative Site, Anniston, Alabama
  - Novartis Investigative Site, Gulf Shores, Alabama
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Chandler, Arizona
  - Novartis Investigative Site, Scottsdale, Arizona
  - Novartis Investigative Site, Buena Park, California
  - Novartis Investigative Site, Norwalk, California
  - Novartis Investigative Site, Westlake Village, California
  - Novartis Investigative Site, Jupiter, Florida
  - Novartis Investigative Site, Largo, Florida
  - Novartis Investigative Site, South Miami, Florida
  - Novartis Investigative Site, Augusta, Georgia
  - Novartis Investigative Site, Decatur, Georgia
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Owensboro, Kentucky
  - Novartis Investigative Site, Metairie, Louisiana
  - Novartis Investigative Site, Troy, Michigan
  - Novartis Investigative Site, Belzoni, Mississippi
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, Picayune, Mississippi
  - Novartis Investigative Site, Missoula, Montana
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Mineola, New York
  - Novartis Investigative Site, New Hyde Park, New York
  - Novartis Investigative Site, Roslyn, New York
  - Novartis Investigative Site, Asheville, North Carolina
  - Novartis Investigative Site, Cary, North Carolina
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, Salisbury, North Carolina
  - Novartis Investigative Site, Shelby, North Carolina
  - Novartis Investigative Site, Wilmington, North Carolina
  - Novartis Investigative Site, Fargo, North Dakota
  - Novartis Investigative Site, Mogadore, Ohio
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Columbia, South Carolina
  - Novartis Investigative Site, Fort Mill, South Carolina
  - Novartis Investigative Site, Greer, South Carolina
  - Novartis Investigative Site, Varnville, South Carolina
  - Novartis Investigative Site, Bristol, Tennessee
  - Novartis Investigative Site, Johnson City, Tennessee
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Bedford, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, League City, Texas
  - Novartis Investigative Site, Bountiful, Utah
  - Novartis Investigative Site, Danville, Virginia
  - Novartis Investigative Site, Midlothian, Virginia
  - Novartis Investigative Site, Newport News, Virginia
  - Novartis Investigative Site, Bellevue, Washington
- Canada (2):
  - Novartis Investigative Site, St. John's, Newfoundland and Labrador
  - Novartis Investigative Site, Sainte-Foy, Quebec
- Germany (5):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Löhne
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Weener
- Lithuania (4):
  - Novartis Investigative Site, Kaunas, LT
  - Novartis Investigative Site, Vilnius, LT
  - Novartis Investigative Site, Klaipėda
  - Novartis Investigative Site, Vilnius

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 68 centers at Canada, Germany, Lithuania, United States from 25-August-2011 (first participant first visit) to 09-May-2013 (last participant last visit).
Pre-assignment Details: A total of 397 participants were randomized in the core study (CACZ885H2361 [NCT01356602]), out of which 232 participants entered the extension study (CACZ885H2361E1 [NCT01431638]).
Groups:
- Canakinumab, Pre-filled Syringes (PFS): Participants received 150 mg subcutaneously (S.C) at randomization and upon new flare. The doses were provided as pre-filled syringes.
- Canakinumab, Lyophilizate (LYO): Participants received 150 mg S.C at randomization and upon new flare. The doses were provided as lyophilized power and had to be reconstituted with water for injection before application.
- Triamcinolone Acetonide: Participants received 40 mg intramuscular (IM) at randomization and upon new flare.
Period: Overall Study
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Started (Core study) | 133 | 132 | 132
Completed Core Study | 124 | 117 | 108
Entered Extension 1 Study | 85 | 71 | 76
Completed (Completed Extension Study) | 67 | 61 | 70
Not Completed | 66 | 71 | 62
Not completed — Adverse Event | 1 | 3 | 1
Not completed — Unsatisfactory therapeutic effect | 2 | 2 | 4
Not completed — Participants condition no longer requires study drug | 0 | 1 | 0
Not completed — Participant withdrew consent | 14 | 5 | 8
Not completed — Lost to Follow-up | 7 | 9 | 7
Not completed — Administrative problems | 1 | 4 | 6
Not completed — Death | 1 | 0 | 0
Not completed — Protocol deviation | 1 | 1 | 4
Not completed — Participants Did not enter extension study from core study | 39 | 46 | 32

BASELINE CHARACTERISTICS:
Population: The analysis was performed in the Randomized Set population defined as all participants who were randomized at least one dose of study drug in the core study (CACZ885H2361 [NCT01356602]).
Groups:
- Total: Total of all reporting groups
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide | Total
Number analyzed (Participants) | 133 | 132 | 132 | 397
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 113 | 104 | 110 | 327
  >= 65-74 years | 15 | 24 | 18 | 57
  >= 75 years | 5 | 4 | 4 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 10 | 34
  Male | 118 | 123 | 122 | 363
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 93 | 93 | 97 | 283
  Black | 35 | 31 | 29 | 95
  Asian | 4 | 4 | 4 | 12
  Native american | 0 | 0 | 0 | 0
  Pacific islander | 0 | 0 | 0 | 0
  Other | 1 | 4 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Reported Adverse Events
Time Frame: From start of the core study (CACZ885H2361 [NCT01356602]) upto end of the current study (48 weeks)
Population: Safety Set consisted of all participants that received study drug in the core study (CACZ885H2361 [NCT01356602]) and had at least one post-baseline safety assessment. The patients with more than one treatment are counted in the Safety Set under those treatment groups as the actual treatments they received. Thus, the number of subjects in the treatment arms are more than the number of randomized subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 133 | 133 | 133
Participants | 78 | 65 | 64

2. Secondary Outcome: Probability of New Gout Flares at End of Study
Description: The Kaplan-Meier estimates of the proportion of participants with first new gout flare, along with the associated 95% confidence intervals using Greenwood's formula were reported. The first new flare was observed either in the core or extension of the study right prior to the switch. The results were reported as Kaplan-Meier estimates.
Time Frame: Up to Day 337
Population: Full Analysis Set (FAS) consisted of all participants randomized in the core study (CACZ885H2361 [NCT01356602]) that had taken at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 131 | 129 | 129
Probability | 65.50 [54.97 to 75.81] | 75.42 [63.82 to 85.57] | 72.95 [62.95 to 82.12]

3. Secondary Outcome: Number of Participant With New Flares
Description: The flare rate was calculated as the number of new flares over the period of observation in years. New flares that occurred before the first study medication dose in the extension 1 study were considered.
Time Frame: up to 36 weeks
Population: FAS consisted of all participants randomized in the core study (CACZ885H2361 [NCT01356602]) that had taken at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 131 | 129 | 129
Participants
  One new flare | 35 | 46 | 36
  Two new flares | 17 | 7 | 26
  Three new flares | 2 | 0 | 8
  Greater (>) than three new flares | 4 | 1 | 3

4. Secondary Outcome: Change From Baseline in Pain Intensity on a 5-point Likert Scale
Description: A Likert scale is a type of scale with a range of responses corresponding to an item such as pain. Participants were advised to score their current pain intensity in the most affected joint of the gouty arthritis flare on a 5-point Likert scale of 1 (None) to 5 (extreme pain), where; 1= none, 2= mild pain, 3= moderate pain, 4= severe pain, or 5= extreme pain (none, mild, moderate, severe, extreme). The higher value presented on the scale was the outcome (high intensity of pain). The respondent selects the best response that indicates the respondent's subjective evaluation of the item. The Last-observation-carried-forward (LOCF) method was used to impute post-dose pain intensity Likert measurements up to 14 days.
Time Frame: Baseline, upto 14 days post-dose
Population: Modified Analysis Set (MAS) consisted of all FAS participants. Here, the number of participants analyzed refer to the participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 42 | 32 | 35
units on a scale | -2.5 (0.86) | -2.3 (0.97) | -2.7 (0.83)

5. Secondary Outcome: Change From Baseline in Pain Intensity in the Most Affected Joint (on a 0-100 mm Visual Analogue Scale [VAS]) Over Time
Description: Patients scored their current pain intensity in the most affected joint of the current gouty arthritis flare on a 0-100 VAS, ranging from no pain (0) to unbearable pain (100). Scores on the 100 mm linear scale were measured to the nearest millimeter from the left.
Time Frame: Baseline, 6, 12, 24, 48, 72 hours post-dose, and Day 4 - 14 post-dose
Population: MAS consisted of all FAS participants. Here, the number of participants analyzed refer to the participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 41 | 32 | 35
units on a scale
  Baseline | 74.2 (14.52) | 75.5 (14.32) | 74.3 (14.44)
  6 hours post-dose | -12.9 (21.03) | -13.0 (17.14) | -10.2 (15.78)
  12 hours post-dose | -23.7 (22.94) | -26.7 (22.09) | -23.4 (19.87)
  24 hours post-dose | -34.9 (24.88) | -36.1 (24.55) | -35.6 (27.09)
  48 hours post-dose | -46.4 (25.31) | -43.8 (24.71) | -51.1 (26.34)
  72 hours post-dose | -55.1 (26.97) | -45.8 (28.74) | -54.7 (30.41)
  4 days post-dose | -55.7 (26.91) | -50.0 (26.39) | -62.0 (23.86)
  5 days post-dose | -59.1 (25.99) | -54.3 (25.43) | -65.2 (23.78)
  6 days post-dose | -61.2 (25.14) | -57.0 (24.27) | -66.0 (23.37)
  7 days post-dose | -62.1 (25.09) | -59.2 (24.32) | -66.6 (22.21)
  8 days post-dose | -59.9 (25.73) | -60.7 (24.07) | -66.8 (22.83)
  9 days post-dose | -63.1 (23.93) | -61.1 (24.34) | -66.7 (23.21)
  10 days post-dose | -63.0 (23.89) | -63.3 (24.31) | -67.9 (22.79)
  11 days post-dose | -62.7 (25.19) | -64.3 (23.53) | -68.7 (22.04)
  12 days post-dose | -63.3 (26.09) | -64.3 (23.91) | -69.4 (20.89)
  13 days post-dose | -65.6 (23.25) | -64.0 (24.47) | -69.6 (20.67)
  14 days post-dose | -64.8 (24.66) | -64.8 (24.15) | -69.8 (21.25)

6. Secondary Outcome: Number of Participants Who Responded for Patient's Global Assessment of Response to Treatment
Description: Participants were advised to make a global assessment of response to treatment using a 5-point Likert scale (1=excellent, 2=good, 3=acceptable, 4=slight, 5=poor).
Time Frame: 48 weeks post-dose
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 72 | 16 | 25
Participants
  Excellent | 50 | 11 | 11
  Good | 17 | 4 | 7
  Acceptable | 2 | 1 | 5
  Slight | 3 | 0 | 1
  Poor | 0 | 0 | 1

7. Secondary Outcome: Number of Participants Responded for Physician's Assessment of Tenderness, Swelling and Erythema of the Most Affected Joint
Description: Tenderness was measured on a 0-3 point scale: no pain, participant states that "there is pain", participant states "there is pain and winces" and participant states "there is pain, winces and withdraws" on palpation or passive movement of the affected study joint. Swelling was measured on a 0 - 3 point scale as follows: 0 = no swelling, 1 = palpable, 2= visible and 3 = bulging beyond the joint margins. Erythema was assessed as present, absent or not assessable.
Time Frame: Baseline, 7 days post-dose
Population: MAS consisted of all FAS participants. Here, the number of participants analyzed refer to the participants evaluable for this outcome measure and at specific category.
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 57 | 49 | 50
Participants
  Tenderness Baseline: No Pain | 0 | 0 | 0
  Tenderness Baseline: Pain | 14 | 6 | 14
  Tenderness Baseline: Pain and winces | 17 | 17 | 20
  Tenderness Baseline: Pain, winces and withdraws | 26 | 26 | 16
  Tenderness 7 days post-dose: No Pain: number analyzed (Participants) | 56 | 49 | 49
  Tenderness 7 days post-dose: No Pain | 42 | 36 | 27
  Tenderness 7 days post-dose: Pain: number analyzed (Participants) | 56 | 49 | 49
  Tenderness 7 days post-dose: Pain | 14 | 12 | 16
  Tenderness 7 days post-dose: Pain, winces: number analyzed (Participants) | 56 | 49 | 49
  Tenderness 7 days post-dose: Pain, winces | 0 | 1 | 5
  Tenderness 7 days post-dose: Pain, winces and withdraws: number analyzed (Participants) | 56 | 49 | 49
  Tenderness 7 days post-dose: Pain, winces and withdraws | 0 | 0 | 1
  Swelling Baseline: No swelling: number analyzed (Participants) | 57 | 49 | 48
  Swelling Baseline: No swelling | 1 | 2 | 4
  Swelling Baseline: Palpable | 9 | 9 | 4
  Swelling Baseline: Visible | 35 | 25 | 27
  Swelling Baseline: Bulging beyond the joint margins | 12 | 13 | 15
  Swelling 7 days post-dose: No swelling: number analyzed (Participants) | 56 | 49 | 49
  Swelling 7 days post-dose: No swelling | 46 | 42 | 38
  Swelling 7 days post-dose: Palpable: number analyzed (Participants) | 56 | 49 | 49
  Swelling 7 days post-dose: Palpable | 8 | 4 | 3
  Swelling 7 days post-dose: Visible: number analyzed (Participants) | 56 | 49 | 49
  Swelling 7 days post-dose: Visible | 2 | 2 | 7
  Swelling 7 days post-dose: Bulging beyond the joint margins: number analyzed (Participants) | 56 | 49 | 49
  Swelling 7 days post-dose: Bulging beyond the joint margins | 0 | 1 | 1
  Erythema Baseline: Absent: number analyzed (Participants) | 56 | 48 | 50
  Erythema Baseline: Absent | 10 | 13 | 15
  Erythema Baseline: Present: number analyzed (Participants) | 56 | 48 | 50
  Erythema Baseline: Present | 46 | 35 | 35
  Erythema 7 days post-dose: Absent: number analyzed (Participants) | 55 | 49 | 49
  Erythema 7 days post-dose: Absent | 51 | 47 | 44
  Erythema 7 days post-dose: Present: number analyzed (Participants) | 55 | 49 | 49
  Erythema 7 days post-dose: Present | 4 | 2 | 5

8. Secondary Outcome: Number of Participants Responded for Physician's Global Assessment of Response to Treatment
Description: The physician made a global assessment of the participant's response to treatment using a 5-point Likert scale: 1=very good, 2=good, 3=fair, 4=poor, 5=very poor.
Time Frame: 7 days post-dose
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
Number analyzed (Participants) | 53 | 49 | 48
Participants
  Very good | 38 | 33 | 32
  Good | 9 | 14 | 13
  Fair | 5 | 2 | 2
  Poor | 1 | 0 | 1
  Very poor | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of the core study (CACZ885H2361 [NCT01356602]) upto end of the current study (48 weeks)
Description: Adverse events were evaluated in the Randomized Set population defined as all participants who were randomized at least one dose of study drug in the core study (CACZ885H2361 [NCT01356602]).
Arm/Group | Canakinumab, Pre-filled Syringes (PFS) | Canakinumab, Lyophilizate (LYO) | Triamcinolone Acetonide
All-Cause Mortality (participants affected / at risk) | 1/133 | 0/132 | 0/132
Serious Adverse Events (participants affected / at risk) | 12/133 | 7/132 | 7/132
Other Adverse Events (participants affected / at risk) | 10/133 | 13/132 | 10/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab, Pre-filled Syringes (PFS) (N=133) | Canakinumab, Lyophilizate (LYO) (N=132) | Triamcinolone Acetonide (N=132)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Drug ineffective (General disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Obstructive uropathy (Renal and urinary disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Aortitis (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab, Pre-filled Syringes (PFS) (N=133) | Canakinumab, Lyophilizate (LYO) (N=132) | Triamcinolone Acetonide (N=132)
Upper respiratory tract infection (Infections and infestations) | 3 | 7 | 1
Hypertension (Vascular disorders) | 7 | 6 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No